CLINICAL TRIAL: NCT00063518
Title: Incidence Rates, Clinical Profile, and Outcomes of Patients With Venous Thromboembolism
Brief Title: Monitoring Trends in Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10387; R01HL070283 (NIH)
Record Dates: First submitted 2003-06-30; First posted 2003-07-01 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Blood Coagulation Disorders; Venous Thromboembolism; Cardiovascular Diseases
MeSH Terms: conditions — Blood Coagulation Disorders; Venous Thromboembolism; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
To describe time trends in the epidemiology of venous thromboembolism.

DETAILED DESCRIPTION:
BACKGROUND:

Venous thromboembolism (VTE) has been estimated to be the third most common cardiovascular disorder. Frequently cited estimates of the incidence of VTE, and its associated outcomes, are based on studies conducted more than a decade ago and only in hospitalized patients. Contemporary data on the magnitude of this disorder, clinical profile of patients affected, acute and long-term outcomes, and use of different treatment strategies are needed given recent advances in diagnostic and therapeutic modalities.

DESIGN NARRATIVE:

The goals of the study are to collect population based data describing trends over time in the epidemiology of VTE including its incidence, management, short and long-term recurrence rates, and mortality. The study will take place in residents of the Worcester, Massachusetts, metropolitan area, (2000 census = 477,800) and will examine changes over time in these and additional endpoints for patients with validated VTE in 1998, 2000 and 2002 with a minimum follow-up of three years. Complementing the community based surveillance of VTE, newly diagnosed cases of VTE occurring in members of the largest Health Maintenance Organization (HMO) in Central Massachusetts between 1998 and 2002 will be identified. This cohort is tracked by an outpatient computer database allowing for the systematic collection of additional data on treatment practices and outcomes occurring outside of the hospital setting. The project will build on the investigators' clinical and epidemiological experience and on data collection methodologies used in the Worcester Deep Vein Thrombosis (DVT) study (1985-1989) and the ongoing Worcester Heart Attack Study. The medical records of Worcester area residents diagnosed with VTE and related diagnostic rubrics will be reviewed and validated according to pre-established diagnostic criteria. Records for additional hospitalizations and death certificates will be reviewed to examine trends in long-term recurrence and survival rates through 2005. The results of this study will provide much needed current reformation about the epidemiology of VTE and provide important data on current diagnostic and therapeutic strategies used in these patients. Implementation of this registry will set the stage for systematic long-term surveillance of this medically important problem.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Spencer, Principal Investigator — University of Massachusetts, Worcester